CLINICAL TRIAL: NCT03555656
Title: Patient Education for the Prevention of Lower Limb Ulcers in Patients With Type 2 Diabetes: Validation of an Educational Intervention Repeated Every Three Months for 2 Years.
Brief Title: Repeated Educational Intervention for the Prevention of Diabetic Foot Ulcers in High-risk Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility analysis suggested termination
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Edoardo Mannucci, Director, Diabetology, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PIEDE2
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repeated educational intervention (Experimental): Repetition every 6 months of a group educational session
  Interventions: Behavioral: Repeated intervention
- Control group (Active Comparator): Initial single group educational session, with no repetition
  Interventions: Behavioral: Single session

INTERVENTIONS:
Behavioral: Repeated intervention — Repetition twice a year of a 2-h group session educating patients at foot hygiene and ulcer prevention
  Arms: Repeated educational intervention
Behavioral: Single session — Single 2-h group session educating patients at foot hygiene and ulcer prevention
  Arms: Control group

SUMMARY:
Following a prior observation that a brief structured group educational intervention is effective for the prevention of diabetic foot ulcers in high-risk patients, but that the efficacy decreases over the time, this study is designed to verify the effect of a repetition of the educational intervention.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Either diabetic neuropathy or previous foot ulcer

Exclusion Criteria:

* Arteriopathy of lower limbs, with ABI<0.8 or needing revascularization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Incidence of foot ulcers | 24 months

SECONDARY OUTCOMES:
Incidence of foot ulcers | 6 months
incidence of foot ulcers | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetologia AOU Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No